CLINICAL TRIAL: NCT00211588
Title: Investigator Initiated Study: Galantamine CR Potential Enhancement of Attentional and Executive Function in Non-Demented Patients With Parkinson's Disease
Brief Title: Galantamine Executive Function in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GAL-EMR-4022
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Parkinson's Disease
Keywords: cognition
MeSH Terms: conditions — Parkinson Disease | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: galantamine

SUMMARY:
The aim of the study is to determine whether galantamine stabilizes or improves thinking abilities in individuals with Parkinson's disease. Individuals included in the study have minor complaints about thinking such as problems with concentration or memory but do not have dementia. This medication has been shown to have a positive effect on stabilizing memory in individuals with Alzheimer's disease. It is FDA approved for use in elderly individuals with Alzheimer's disease. It is hypothesized that galantamine will stabilize or improve executive and attentional functions in individuals with Parkinson's.

DETAILED DESCRIPTION:
While several cholinesterase inhibitors have effectiveness in Alzheimer's disease (AD), galantamine is unique since it has a dual mode of action: inhibition of acetylcholinesterase and modulation of nicotinic acetylcholine receptors.As Parkinson's disease (PD) impacts frontal systems, executive cognition rather than memory function (mediated by medial temporal) would be the targeted area for potential improvement. This single center, double blind, placebo controlled study compares a group of PD patients treated with galantamine to a group of PD patients who are not treated with this medication on a series of cognitive tasks that examine attention and executive control.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease

Exclusion Criteria:

* dementia, depression, cardiac disease, gastrointestinal disease

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2004-06; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Improvement on cognitive measures | 16 weeks

SECONDARY OUTCOMES:
No worsening of PD symptoms | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Friedman, M.D., Principal Investigator — NeuroHealth; Janet Grace, Ph.D., Study Director — Memorial Hospital of RI
Locations (1):
- Memorial Hospital of RI, Pawtucket, Rhode Island, United States

REFERENCES:
- [Derived] Buelow MT, Amick MM, Queller S, Stout JC, Friedman JH, Grace J. Feasibility of use of probabilistic reversal learning and serial reaction time tasks in clinical trials of Parkinson's disease. Parkinsonism Relat Disord. 2015 Aug;21(8):894-8. doi: 10.1016/j.parkreldis.2015.05.019. Epub 2015 May 27. PMID 26040709